CLINICAL TRIAL: NCT01843725
Title: Modulation of Metabolic Index in Tailoring Treatment of Incurable Metastatic ColoRectal Cancer (CRC) Program 1.
Brief Title: Phase 1 Study Testing the Combination of Aflibercept and Capecitabine in Metastatic Digestive and Breast Cancers
Acronym: MOMENTUM1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mom1-AD12; 2012-005169-11 (EudraCT Number)
Record Dates: First submitted 2013-04-25; First posted 2013-05-01 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Colorectal Cancers; Metastatic Gastric Cancers; Metastatic Oesophageal Cancers; Metastatic Pancreatic Cancers; Metastatic Biliary Cancers; Metastatic Breast Cancers
Keywords: breast cancer; digestive cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms; Breast Neoplasms; Gastrointestinal Neoplasms | interventions — Capecitabine; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronomic arm (Experimental): capecitabine 1100 to 1600 mg/m2/day orally in association with aflibercept 6mg/kg intravenous every 3 weeks
  Interventions: Drug: capecitabine; Drug: aflibercept
- Intermittent arm (Experimental): capecitabine 1700 to 2500 mg/m2/day orally 2 weeks out of 3 and aflibercept 6mg/kg intravenous every 3 weeks
  Interventions: Drug: aflibercept; Drug: Capecitabine

INTERVENTIONS:
Drug: capecitabine — escalation dose of capecitabine continuously
  Other Names: Xeloda
  Arms: Metronomic arm
Drug: aflibercept — Intravenous 6mg/kg every 3 weeks
  Other Names: Zaltrap
Drug: Capecitabine — dose escalation, from 1700 to 2500mg/m2/day 2 weeks out of 3
  Other Names: Xeloda
  Arms: Intermittent arm

SUMMARY:
Prospective non randomized, non-comparative, dose escalation, two arms open phase I trial to assess the safety and tolerability of capecitabine given in combination with aflibercept in patients with measurable or evaluable, chemorefractory digestive tumors or breast tumors in terms of the Maximum Tolerated Dose (MTD) and the Dose-Limiting Toxicities (DLTs), To establish the Recommended Phase II Dose (RP2D) of capecitabine in combination with Aflibercept.

DETAILED DESCRIPTION:
Aflibercept has been found to be active with a broad pharmacological index against early and advanced stage disease in a variety of preclinical solid tumor models including sarcomas, and ovarian, prostate, mammary, colon, and gastric carcinomas either as a single agent or in combination with cytotoxic agents.

Metronomic chemotherapy, namely administration of continuous low-dose chemotherapy at close, regular intervals, with no prolonged drug-free interruptions, bases its rationale on the fact that virtually all classes of cancer chemotherapeutic drugs are designed to damage DNA or disrupt microtubules of dividing cells. Endothelial cell division takes place during new blood vessel formation, including tumour angiogenesis. Frequent administration of most cytotoxic agents at low doses is thought to increase their putative antiangiogenic activity.

This strategy lowers the toxicity and theoretically the risk of emergence of drug-resistant tumour cells compared to classic maximum tolerated dose (MTD)-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed digestive or breast cancer that is metastatic or unresectable, for which no curative measures are possible, and chemorefractory to all known medications in the respective fields.
* Age ≥ 18 years.
* Life expectancy of greater than 12 weeks.
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 1.
* Normal organ and marrow function as defined below:

  * Leukocytes > 3,000/microLiter (mcL)
  * Hb>10g/mcL
  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * Total bilirubin within 2 × institutional upper limit of normal
  * AST (aspartate amino transferase)/ALT (alanine amino transferase)/ALKP (Alkaline Phosphatase) levels < 5 × institutional upper limit of normal for liver metastases, < 2.5 ULN (Upper Limit of Normal) in case of no liver metastases
  * Creatinine within 2 × institutional upper limit of normal or creatinine clearance > 35 mL/min
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Signed written informed consent (approved by an Independent Ethics Committee (IEC)) obtained prior to any study specific baseline procedures.

Exclusion Criteria:

* Patients with malabsorption or dysfunctional GI tract.
* Participants who have had chemotherapy or radiotherapy (except limited radiotherapy for bone metastasis for instance) within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants should not receive any other experimental agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

  * History of cardiovascular ischemic disease or cerebrovascular incident within the last six months, NYHA class III and IV congestive heart failure.
  * Intolerance to atropine sulfate or loperamide
  * Known dihydropyrimidine dehydrogenase deficiency
  * Treatment with CYP3A4 inducers unless discontinued > 7 days prior to randomization
  * Any of the following in 3 months prior to inclusion: grade 3-4 gastrointestinal bleeding (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, or diverticulitis.
* Major surgery within 6 weeks.
* Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women, lactation or refusal to use adequate contraceptive measures (hormonal or barrier method of birth control, abstinence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and the recommended phase II dose of capecitabine in association with aflibercept | The time point of the first toxicity evaluation would be the end of the first cycle (3 weeks)
  To assess the safety and tolerability of capecitabine given in combination with aflibercept in patients with measurable or evaluable, chemorefractory digestive tumors or breast tumors in terms of the Maximum Tolerated Dose (MTD), the Dose-Limiting Toxicities (DLTs), and to determine the Recommended Phase II Dose (RP2D) of capecitabine in combination with aflibercept.

SECONDARY OUTCOMES:
The secondary endpoint is preliminary data on efficacy, and this will be evaluated using CT scan or MRI using RECIST (Response Evaluation Criteria in Solid Tumors) v1.1 | after 2 cycles (6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Hendlisz, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

REFERENCES:
- [Derived] Camera S, Deleporte A, Bregni G, Trevisi E, Pretta A, Telli TA, Polastro L, Gombos A, Kayumba A, Ameye L, Piccart-Gebhart M, Awada A, Sclafani F, Hendlisz A. MOMENTUM: A Phase I Trial Investigating 2 Schedules of Capecitabine With Aflibercept in Patients With Gastrointestinal and Breast Cancer. Clin Colorectal Cancer. 2020 Dec;19(4):311-318.e1. doi: 10.1016/j.clcc.2020.05.007. Epub 2020 May 29. PMID 32631787